CLINICAL TRIAL: NCT07029282
Title: A Phase III Double-Blind, Adaptive Randomized Trial of Antenatal MMSPlus Versus UNIMAPP MMS and Postnatal MMSPlus Versus UNIMAPP MMS or IFA to Improve Infant Birth Outcomes and Growth at 6 Months
Brief Title: The MOM-CARE Trial : Evaluating Antenatal and Postnatal MMSPlus for Improved Infant Birth and Growth Outcomes
Acronym: MOM-CARE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Vital Pakistan Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-10733-31927
Record Dates: First submitted 2025-05-23; First posted 2025-06-19 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Newborn Health; Multiple Micronutrient Deficiencies During Pregnancy; Nutrition During Pregnancy; Adaptive Trial; Postnatal Growth; Neurodevelopment Outcome
Keywords: Antenatal Phase; Postnatal Phase; Micro Nutrient Supplementation; Infant Growth

STUDY DESIGN:
Intervention Model Description: During the antenatal phase, participants will be randomized into one of two arms (MMS vs MMS Plus). However during the postnatal phase, those same participants will be re-randomized into three arms (MMS vs MMS Plus vs IFA).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MMS (Active Comparator): Once daily dose of MMS sachet + Standard ANC and nutrition counseling
  Interventions: Dietary Supplement: MMS
- IFA (Active Comparator): Once daily dose of IFA sachet + Standard postnatal care (PNC) and nutrition counseling
  Interventions: Dietary Supplement: IFA
- MMS Plus (Experimental): One daily sachet of MMS PLUS + Standard ANC and nutrition counseling
  Interventions: Drug: MMS Plus

INTERVENTIONS:
Dietary Supplement: MMS — Pregnant women in this arm will receive 6gms of MMS (UNIMAPP MMS) in a ready to use sachet form which includes 15 nutrients.
  Other Names: UNIMAPP MMS
  Arms: MMS
Drug: MMS Plus — Pregnant women in this arm will receive 6gms of MMS Plus in a ready to use sachet form which includes 18 nutrients.
  Arms: MMS Plus
Dietary Supplement: IFA — Pregnant women in this arm will receive 6gms of IFA (Iron/Folic Acid) in a ready to use sachet form which includes 2 nutrients.
  Arms: IFA

SUMMARY:
This clinical trial aims to learn if MMS Plus improves infant health compared to standard MMS during pregnancy and the postnatal period in women living in peri-urban areas of Karachi, Pakistan. It will also evaluate how MMS Plus affects infant growth during the first 6 months of life.

The main questions it aims to answer are:

1. Does MMS Plus during pregnancy reduce the risk of poor infant outcomes compared to standard MMS, as measured on a 5-point ordinal scale ranging from perinatal mortality to term birth with appropriate, small, or large-for-gestational-age infants?
2. Does postnatal MMS Plus improve infant length velocity at 6 months of age among exclusively breastfed infants compared to standard MMS and iron/folic acid (IFA) supplementation?

Researchers will compare:

1. MMS Plus versus standard MMS during pregnancy (antenatal phase)
2. MMS Plus versus standard MMS versus IFA after birth (postnatal phase)

Participants will:

1. Be randomly assigned to receive either MMS Plus or standard MMS during pregnancy
2. Be re-randomized after delivery to receive either MMS Plus, standard MMS, or IFA supplements during the postnatal period
3. Receive supplements under double-blind conditions
4. Be followed through childbirth and until the infant is 6 months of age
5. Attend regular clinic visits for health monitoring, infant assessments, and data collection.

This phase III adaptive randomized controlled trial will occur in three peri-urban catchment areas of Karachi, Pakistan.

DETAILED DESCRIPTION:
This is a two-phase, Phase III double-blind, adaptive randomized controlled trial designed to evaluate the effects of enhanced multiple micronutrient supplementation (MMS Plus) compared to standard UNIMMAP MMS and iron/folic acid (IFA) supplementation on maternal and infant health outcomes in peri-urban Karachi, Pakistan. The trial is being conducted by The Aga Khan University and is funded by the Bill Gates Foundation.

Study Phases and Design:

Antenatal Phase:

Pregnant women between 8-14 weeks of gestation will be enrolled and randomized (1:1) into one of two arms:

MMS Plus (enhanced formulation) Standard MMS (UNIMMAP formulation)

Both groups will also receive standard antenatal care (ANC) and nutrition counseling. The primary endpoint is a composite 5-point ordinal scale of infant health at 28 days post-birth, which includes perinatal mortality and growth-for-gestational-age outcomes - Small for gestational age (SGA), Appropriate for Gestational Age (AGA) and Large for Gestational Age (LGA), along with preterm or term. The trial employs a Bayesian adaptive design, with interim analyses beginning after 500 participants have birth outcomes, and subsequent evaluations every 250 outcomes. The design allows early stopping for superiority or continuation based on posterior probabilities.

Postnatal Phase:

Women with live births will be re-randomised (1:1:1) within one week postpartum into one of three arms:

MMS Plus Standard MMS IFA (standard care)

All groups receive standard postnatal care and nutrition counselling. The primary endpoint is infant length velocity (cm/month) at 6 months among exclusively breastfed infants. Secondary outcomes include additional anthropometric measures and neurodevelopmental assessments. Adaptive analyses in this phase also begin after 500 infants have outcome data.

Interventions:

MMS Plus includes 22 micronutrients with additional components: choline (450 mg), DHA (200 mg), calcium (500 mg), and a higher dose of nicotinamide (118 mg NE).

Standard MMS follows the UNIMMAP formulation with 15 micronutrients. IFA includes 60 mg of iron and 400 mcg folic acid.

All supplements are administered daily via single-dose sachets, indistinguishable in packaging and taste to preserve blinding. Products are manufactured by Remington Pharma.

Setting and Recruitment:

The trial is implemented through the Clinical Trials Unit (CTU) of Aga Khan University. Recruitment will occur in three peri-urban catchment communities: Ali Akbar Shah Goth (AG), Bhains Colony (BH), and Qayyumabad (QB). Two sites (AG and BH) are located in District Malir and one (QB) in District East. These communities have been selected due to high burdens of maternal undernutrition and established surveillance systems through the Integrated Research Platform (IRP).

Pregnant women will be recruited during Antenatal Care (ANC) visits and confirmed eligible via ultrasound. Postnatal re-randomization occurs for women with eligible live-born infants. Follow-up includes scheduled home and clinic visits until 6 months postpartum. Participants will receive all clinical services and transportation free of charge.

Data Management and Monitoring:

Data will be collected using a digital platform developed on OpenSRP, enabling longitudinal tracking of mother-child dyads. Unique IDs link all clinical encounters and supplement adherence records. Data quality assurance includes weekly field audits, double-entry verification, and remote monitoring by the trial coordination team.

A Data Safety Monitoring Board (DSMB) will review interim results and safety data. Trial governance includes a Trial Management Group (TMG) and an independent Trial Steering Committee. All adverse events will be reported following institutional and national regulatory guidelines.

Scientific Rationale:

Despite global efforts to improve maternal and infant nutrition, Pakistan continues to report high levels of maternal anaemia, low birth weight, and childhood stunting. While MMS is being piloted for national scale-up, the evidence base for extended formulations remains limited, especially regarding postnatal supplementation. MMS Plus is hypothesised to offer superior outcomes due to its inclusion of neurodevelopmentally and metabolically relevant nutrients (choline, DHA, calcium, and high-dose nicotinamide). These additions are based on recent findings from the MUMTA trial and other global data highlighting their role in fetal brain development, infant growth, and maternal health.

This trial addresses critical knowledge gaps in the timing (antenatal vs. postnatal), formulation, and impact of micronutrient interventions, using robust adaptive methodologies to optimise power, efficiency, and ethical participant exposure.

ELIGIBILITY:
Antenatal Phase::

Inclusion Criteria:

* Gestational age confirmed by ultrasound to be 8-14 weeks
* Singleton and viable fetus on ultrasound
* A resident of the catchment area for at least the last six months
* Plans to stay within the catchment area during the pregnancy duration, during delivery and after birth of the baby.
* Has provided voluntary written informed consent

Exclusion Criteria:

* Women with known allergies or intolerance to any components of the MMS or MMS PLUS being studied
* Women with pre-existing health conditions such as history of uncontrolled diabetes and hypertension or other chronic illnesses
* Substance abuse, such as recreational drugs or smoking tobacco. Women chewing tobacco will not be excluded.

Postnatal Phase::

Inclusion Criteria:

* Birth weight available within 72 hours
* Intention to breastfeed for 6 months
* Resides in the study area for the duration of the trial
* Has provided voluntary written informed consent

Exclusion Criteria:

* Congenital anomalies, birth defects, or severe neonatal complications
* Infants who are already receiving supplemental formula feeding or other nutritional supplements (except pre-lacteal feeding, vitamins, and medications)
* Infants whose mothers have conditions that significantly affect breastfeeding, such as severe postpartum depression, insufficient milk supply, or maternal use of medications that contraindicate breastfeeding

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Antenatal Phase: Composite Infant Health Score at 28 Days Post-Birth | 28 days after birth
  Infant health will be assessed using a 5-point ordinal categorical scale, defined as follows:
  Stillbirth, miscarriage, or early neonatal death (0-6 days); Preterm birth with Small for Gestational Age (SGA) infant; Preterm birth with Appropriate or Large for Gestational Age (AGA or LGA) infant; Term birth with SGA infant; Term birth with AGA or LGA infant Method of Aggregation: Proportion of participants in each outcome category Analysis Metric: Ordinal regression (e.g., Bayesian cumulative logistic regression)
Postnatal Phase: Infant linear growth velocity at 6 months | Birth to 6 months
  Infant linear growth velocity, calculated as:
  Length Velocity (cm/month) = Length at 6 months - Length at birth / Age in days / 30.4 Only infants exclusively/predominantly breastfed through 6 months will be included in this analysis.
  Method of Aggregation: Mean length velocity per intervention group Analysis Metric: Continuous variable; analysed using ANOVA or regression models with pairwise comparisons

SECONDARY OUTCOMES:
Gestational Weight Gain (GWG) | At birth
  Change in maternal weight during pregnancy, measured in kilograms (kg) from baseline (enrollment) to the time of delivery.
  Gestational weight gain will be reported both as:
  Absolute weight gain (kg) Z-scores and percentiles, adjusted for gestational age, based on WHO or INTERGROWTH standards
  Greater weight gain within recommended ranges is considered indicative of improved maternal nutritional status and better fetal outcomes.
Intrauterine Growth Restriction (IUGR) | GA 20 and 32 weeks
  Episodes of IUGR measured at two timepoints during antenatal phase measured through ultrasound to assess growth of fetus in relation to weight and size
Gestational age at birth | Within 72 hours of birth
  Gestational age at birth, measured in completed weeks, will be assessed using first-trimester ultrasound dating (8-14 weeks gestation).
  Higher gestational age indicates a better outcome in terms of fetal maturity and reduced risk of neonatal complications.
  Method of aggregation: Mean gestational age (weeks); proportion of births in each gestational age category (preterm, term, post-term)
Birth Weight (gm) | Within 72 hours of birth
  Weight of the newborn assess in gram to assess the difference between the arms
Birth length (cm) | within 72 hours of birth
  Length of the newborn assess in cm to assess the difference between the arms
Head circumference (cm) | within 72 hours of birth
  Head circumference of the newborn assess in cm to assess the difference between the arms
Infant MUAC (cm) | within 72 hours of birth
  Infant MUAC at birth of the newborn assess in cm to assess the difference between the arms
Neonatal Mortality | within the first 28 days of life
  Neonatal mortality to assess the difference between arms
Infant weight velocity | 1, 2, 4, 6, 12, 24 months of life
  Mean difference in growth velocity of >0.4 gram/kg/day to look at comparisons between multiple arms
Length-for-age z-score (LAZ) | 2, 4, 6, 12, 24 months of life
  Mean difference in LAZ >0.5 to look at comparisons between multiple arms
Weight-for-age z-score (WAZ) | 2, 4, 6, 12, 24 months of life
  Mean difference in WAZ of >0.5 to look at comparisons between multiple arms
Stunting, wasting and underweight Stunting <-2 LAZ ( Length for age Z) scores; Wasting <-2 WHZ (Weight for height Z) scores; underweight <-2WAZ (Weight for age Z) scores | 2, 4, 6, 12, 24 months of life
  Mean difference in LAZ, WHZ and WAZ scores to look at comparison between multiple arms
Global Scale for Early Development (GSED) Assessment | 6, 12 and 24 months of life
  Neurodevelopmental functioning will be assessed using the Global Scales for Early Development (GSED), a standardised instrument developed by the World Health Organisation to measure early child development across cognitive, motor, language, and socio-emotional domains.
  The GSED yields a Developmental Score (D-score), which is a continuous score derived from observed developmental milestones.
  Minimum Value: ~30 (varies slightly based on age and item completion)
  Maximum Value: ~80
  Interpretation: Higher scores indicate better neurodevelopmental status
  Scores will be analysed as continuous variables and categorised into:
  "On track"
  "At risk"
  "Developmental delay" based on GSED normative thresholds for age.
Infant Brain Morphology and Volume (MRI Assessment Using Hyperfine Portable MRI) | 6, 12 and 24 months of life
  Infants enrolled in the postnatal phase will undergo brain imaging using the Hyperfine Swoop™ portable MRI system to assess brain morphology and total and regional brain volumes.
  Imaging will be conducted at 6, 12, and 24 months of age.
  Brain volume will be quantified in cubic centimetres (cc) for total brain, grey matter, white matter, and selected regions of interest (e.g., hippocampus, cerebellum).
  Morphological features (e.g., sulcal/gyral patterns, ventricular size, myelination status) will be qualitatively described and coded using standardised radiological criteria.
  Higher volumes and normal morphology are indicative of better neurodevelopmental outcomes.

OTHER OUTCOMES:
Maternal weight | 1, 2, 4, 6, 12, 24 months of life
  Maternal body weight, measured in kilograms (kg), will be assessed after delivery to evaluate maternal nutritional status following supplementation during the postnatal phase. Weight will be measured using calibrated digital scales under standardized conditions.
  Higher weight (within normal postpartum range) indicates better nutritional recovery and health status.
Maternal MUAC (cm) | 1, 2, 4, 6, 12, 24 months of life
  Mean difference of MUAC in cm to look at comparison between multiple arms
Maternal morbidity | Every ANC visit and within 72 hours of birth
  Episodes of maternal morbidities such as preeclampsia, gestational diabetes mellitus, hypertensive disorders in between the arms

CONTACTS AND LOCATIONS:
Overall Officials: Fyezah Jehan, MBBS; MSc, Principal Investigator — Aga Khan University
Locations (1):
- Peri-Urban Slums of Karachi (Ali Akber Shah, Bhains Colony), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
It will most likely be shared, but it has not been decided how, yet.

REFERENCES:
- [Background] Amoroso L. Post-2015 Agenda and Sustainable Development Goals: Where Are We Now? Global Opportunities to Address Malnutrition in all Its Forms, Including Hidden Hunger. World Rev Nutr Diet. 2017;118:45-56. doi: 10.1159/000484334. Epub 2018 Apr 13. PMID 33503779
- [Background] GNR. The state of global nutrition. Development Initiatives Bristol (UK); 2021
- [Background] UNICEF. National Nutrition Survey 2018. Key Findings Report Ministry of Health Services, Nutrition Wing, Regulation and Coordination, Government of Pakistan, Pakistan. 2019
- [Background] WHO Recommendations on Antenatal Care for a Positive Pregnancy Experience. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK409108/ PMID 28079998
- [Background] Bourassa MW, Osendarp SJM, Adu-Afarwuah S, Ahmed S, Ajello C, Bergeron G, Black R, Christian P, Cousens S, de Pee S, Dewey KG, Arifeen SE, Engle-Stone R, Fleet A, Gernand AD, Hoddinott J, Klemm R, Kraemer K, Kupka R, McLean E, Moore SE, Neufeld LM, Persson LA, Rasmussen KM, Shankar AH, Smith E, Sudfeld CR, Udomkesmalee E, Vosti SA. Review of the evidence regarding the use of antenatal multiple micronutrient supplementation in low- and middle-income countries. Ann N Y Acad Sci. 2019 May;1444(1):6-21. doi: 10.1111/nyas.14121. Epub 2019 May 27. PMID 31134643
- [Background] Keats EC, Haider BA, Tam E, Bhutta ZA. Multiple-micronutrient supplementation for women during pregnancy. Cochrane Database Syst Rev. 2019 Mar 14;3(3):CD004905. doi: 10.1002/14651858.CD004905.pub6. PMID 30873598
- See also: WHO, Malnutrition, 2021 — https://www.who.int/news-room/fact-sheets/detail/malnutrition